CLINICAL TRIAL: NCT03945981
Title: A Phase 3b Multi-center, Open Label, Single Arm, 52-week Study, Evaluating the Feasibility, Efficacy and Safety of Rapid Test and Treat Intervention in Newly Diagnosed HIV-1 Infected Adults Using a Fixed Dose Combination of Dolutegravir Plus Lamivudine (DOVATO) as a First Line Regimen
Brief Title: Rapid Test and Treat Dolutegravir Plus Lamivudine Study in Newly Diagnosed Human Immunodeficiency Virus (HIV)-1 Infected Adults
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: ViiV Healthcare (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 212355
Record Dates: First submitted 2019-05-08; First posted 2019-05-10 (Actual); Results first posted 2021-04-28 (Actual); Last update posted 2021-10-21 (Actual); Status verified 2021-09

CONDITIONS: HIV Infections
Keywords: GSK3515864, dolutegravir, Dovato, lamivudine, 3TC, HIV-1, Test and Treat
MeSH Terms: conditions — HIV Infections | interventions — dolutegravir

STUDY DESIGN:
Intervention Model Description: Participants will receive 50 mg DTG + 300 mg 3TC FDC, participants will administer one tablet once daily (OD) orally with or without food.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- Participants receiving Dolutegravir + Lamivudine FDC (Experimental): Participants will receive DTG 50mg and 3TC 300 mg FDC tablet orally once daily (OD) with or without food
  Interventions: Drug: Dolutegravir + Lamivudine FDC

INTERVENTIONS:
Drug: Dolutegravir + Lamivudine FDC — Dolutegravir + Lamivudine FDC is available as white oval film-coated tablets which are packed in high density polyethylene (HDPE) bottles with induction seals and child-resistant closures. Each 60 milliliter (mL) bottle contains 30 tablets

SUMMARY:
Early initiation of antiretroviral therapy (ART) reduces morbidity and mortality for individuals infected with HIV. Suppressing viral replication with ART also reduces the potential for transmission of HIV. Hence, ART is recommended for all persons with HIV viremia regardless of cluster of differentiation 4 (CD4) count. This is an open-label single arm which will evaluate the feasibility, efficacy and safety using a fixed dose combination (FDC) of Dolutegravir (DTG) plus Lamivudine (3TC) as a first line regimen of a rapid Test and Treat model of care over 48 weeks. Participants with new and confirmed diagnosed HIV-1 who are willing to start study treatment immediately following diagnosis will receive 50 milligram (mg) DTG + 300 (mg) 3TC FDC as first line therapy without waiting for screening laboratory results, at the Screening/Day 1 Visit. The total duration for the study will be 52 weeks and 4 weeks of follow up period if required. This study will be conducted in United States (US) with approximately 120 participants.

ELIGIBILITY:
Inclusion Criteria:

* Eligible participants must be able to understand and comply with protocol requirements, instructions, and restrictions.
* Eligible participants must be likely to complete the study as planned.
* Eligible participants must be considered appropriate candidates for participation in an investigative clinical trial with oral medication (e.g. no active problematic substance abuse, acute major organ disease, or potential long-term work assignments out of the country).
* Participant must be more than or equal to 18 at the time of signing the informed consent.
* Participants must have a new and confirmed diagnosis of HIV-1 infection and are willing to initiate ART immediately (or, for those participants referred from another site, within 14 days of initial diagnosis at the external clinic/testing center).
* Participant must have an initial positive rapid HIV test and participant has a second positive confirmatory rapid HIV test, using a test kit from a different manufacturer than the first test or participant has been identified as HIV-1 infected using an FDA-approved 4th generation assay antigen/antibody combination immunoassay or 3rd generation immunoassay that detects and differentiates HIV-1 and HIV-2 antibodies; participant has a confirmatory HIV western blot or an HIV-1 RNA or participant has a positive FDA-approved 4th generation assay and a positive 3rd generation immunoassay that detects and differentiates HIV-1 and HIV-2 antibodies.
* Antiretroviral-naïve. Participants who received HIV post-exposure prophylaxis (PEP) or pre-exposure prophylaxis (PrEP) in the past are allowed as long as the last PEP/PrEP dose was more than 6 months from HIV diagnosis or there is documented HIV seronegativity at least 2 months after the last prophylactic dose and prior to the date of HIV diagnosis.
* Male and/or female participants.
* Participants who are female at birth are eligible to participate if at least one of the following conditions applies: Not pregnant [as confirmed by a negative urine human chorionic gonadotropin (hCG) test at Screening/Day 1.
* Pregnant and post the first trimester (the physician and patient should decide whether enrolling in this study is in the participants best interest during the consent process)
* Not a participant of childbearing potential (POCBP) or a POCBP agrees to follow the contraceptive guidance, is currently taking hormonal contraceptives and continues for at least 2 weeks after the last dose of study medication. Participants who are female at birth and who are in the following categories are not considered POCBP, premenarchal, premenopausal female with one of the following: documented hysterectomy, documented bilateral salpingectomy, documented bilateral oophorectomy or postmenopausal, a postmenopausal state is defined as no menses for 12 months without an alternative medical cause; a high follicle stimulating hormone (FSH) level in the postmenopausal range may be used to confirm a postmenopausal state in participants who are female at birth and not using hormonal contraception or hormonal replacement therapy (HRT); participants who are female at birth on HRT and whose menopausal status is in doubt will be required to use one of the non-hormonal highly effective contraception methods if they wish to continue their HRT during the study.
* Participants who are capable of giving signed informed consent which includes compliance with the requirements and restrictions listed in the informed consent form (ICF) and in this protocol.

Exclusion Criteria:

* Participants who are breastfeeding, plan to become pregnant or breastfeed during the study.
* Participants who are in their first trimester of pregnancy.
* HIV-1 drug resistance genotype test results are known prior to Screening/Day 1.
* Any evidence of an active Centers for Disease Control and Prevention (CDC) Stage 3 disease except for esophageal candidiasis and cutaneous Kaposi's sarcoma not requiring systemic therapy.
* Participants with known or suspected Hepatitis B infection.
* Participants with known or suspected severe hepatic impairment or unstable liver disease (as defined by the presence of ascites, encephalopathy, coagulopathy, hypoalbuminemia, esophageal or gastric varices, or persistent jaundice), cirrhosis, known biliary abnormalities (with the exception of Gilbert's syndrome or asymptomatic gallstones).
* Participants with known moderate to severe renal impairment (creatinine clearance less than 30ml/minute per 1.73 square meter);
* Participant with ongoing malignancy other than basal cell carcinoma, or resected, non-invasive cutaneous squamous cell carcinoma, or cervical, anal or penile intraepithelial neoplasia; other localized malignancies require agreement between the investigator and the Study Medical Monitor for inclusion of the participant.
* Participants who in the investigator's judgment, poses a significant suicidality risk.
* Participants with any pre-existing physical or mental condition which, in the opinion of the Investigator, may interfere with the participant's ability to comply with the dosing schedule and/or protocol evaluations or which may compromise the safety of the participant.
* Participants with substance abuse disorders or social restraints that the Investigator considers to be possible deterrents to successful initiation of ART.
* Participants with history or presence of allergy or intolerance to the study drugs or their components.
* Participants with treatment with any of the following agents within 28 days of the first dose of study treatment, radiation therapy, cytotoxic chemotherapeutic agents, any systemic immune suppressant.
* Participants receiving any prohibited medication and who are unwilling or unable to switch to an alternate medication.
* Exposure to an experimental drug or experimental vaccine within either 28 days, 5 half-lives of the test agent, or twice the duration of the biological effect of the test agent, whichever is longer, prior to the first dose of study treatment.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 131 (Actual)
Dates: Start 2019-07-02 (Actual); Primary Completion 2020-04-29 (Actual); Study Completion 2020-10-20 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: GSK Clinical Trials, Study Director — ViiV Healthcare
Locations (15):
- United States (15):
  - GSK Investigational Site, Birmingham, Alabama
  - GSK Investigational Site, Los Angeles, California
  - GSK Investigational Site, Palm Springs, California
  - GSK Investigational Site, Ft. Pierce, Florida
  - GSK Investigational Site, Miami, Florida
  - GSK Investigational Site, Oakland Park, Florida
  - GSK Investigational Site, Orlando, Florida
  - GSK Investigational Site, Decatur, Georgia
  - GSK Investigational Site, Savannah, Georgia
  - GSK Investigational Site, Minneapolis, Minnesota
  - GSK Investigational Site, St Louis, Missouri
  - GSK Investigational Site, Huntersville, North Carolina
  - GSK Investigational Site, Austin, Texas
  - GSK Investigational Site, Bellaire, Texas
  - GSK Investigational Site, Dallas, Texas

IPD SHARING:
Plan to Share IPD: Yes
IPD for this study will be made available via the Clinical Study Data Request site.
Supporting Information: Study Protocol, SAP, ICF, CSR
Time Frame: IPD will be made available within 6 months of publishing the results of the primary endpoints of the study.
Access Criteria: Access is provided after a research proposal is submitted and has received approval from the Independent Review Panel and after a Data Sharing Agreement is in place. Access is provided for an initial period of 12 months but an extension can be granted, when justified, for up to another 12 months.
URL: http://clinicalstudydatarequest.com

REFERENCES:
- [Background] Rolle CP, Berhe M, Singh T, Ortiz R, Wurapa A, Ramgopal M, Leone PA, Matthews JE, Dalessandro M, Underwood MR, Angelis K, Wynne BR, Merrill D, Nguyen C, van Wyk J, Zolopa AR. Dolutegravir/lamivudine as a first-line regimen in a test-and-treat setting for newly diagnosed people living with HIV. AIDS. 2021 Oct 1;35(12):1957-1965. doi: 10.1097/QAD.0000000000002979. PMID 34115650
- [Derived] Rolle CP, Arribas JR, Ortiz R, Underwood M, Parry CM, Grove R, DiMondi VP, Jones B, Kisare M. Efficacy and Safety Outcomes in Adults Initiating Dolutegravir/Lamivudine With High Viral Load in the GEMINI-1/-2 and STAT Trials. Open Forum Infect Dis. 2025 Mar 7;12(3):ofaf135. doi: 10.1093/ofid/ofaf135. eCollection 2025 Mar. PMID 40134635

RESULTS

PARTICIPANT FLOW:
Recruitment Details: This was an open-label single arm study to evaluate the feasibility, efficacy and safety of a rapid Test and Treat intervention in newly diagnosed human immunodeficiency viruses (HIV)-1 infected adults using a fixed dose combination of dolutegravir (DTG) plus lamivudine (3TC) as a first line regimen.
Pre-assignment Details: A total of 133 participants were screened and 131 participants were enrolled in the study.
Groups:
- DTG Plus 3TC: Participants received DTG 50 milligram (mg) and 3TC 300 mg fixed dose combination tablet orally once daily with or without food.
Period: Overall Study
Arm/Group | DTG Plus 3TC
Started | 131
Completed | 108
Not Completed | 23
Not completed — Lost to Follow-up | 12
Not completed — Physician Decision | 4
Not completed — Withdrawal by Subject | 6
Not completed — Protocol Violation | 1

BASELINE CHARACTERISTICS:
Arm/Group | DTG Plus 3TC
Number analyzed (Participants) | 131
Age, Continuous [Mean (Standard Deviation); unit: Years] | 34.6 (11.46)
Sex/Gender, Customized [Number; unit: Participants]
  Male | 120
  Female | 10
  Transgender Female | 1
Race/Ethnicity, Customized [Number; unit: Participants]
  American (Amer.) Indian(Ind.)orAlaska(Ala.)Native | 1
  Central/South Asian Heritage | 2
  African American/African (Afr.) Heritage (Her.) | 61
  Native Hawaiian or other Pacific Islander | 1
  White/Caucasian/European Heritage | 65
  Afr.Amer./Afr. Her. and Amer. Ind. or Ala. Native | 1

OUTCOME MEASURES:

1. Primary Outcome: Percentage of Participants With Plasma Human Immunodeficiency Virus Type 1 (HIV-1) Ribonucleic Acid (RNA) <50 Copies/Milliliter (c/mL) Regardless of Antiretroviral Therapy (ART) Regimen at Week 24 by ITT-E Missing = Failure Analysis
Description: Participants were classified as "HIV-1 RNA <50 c/mL" using an ITT-E missing = Failure analysis. Participants were classified as 'HIV-1 RNA < 50 c/mL' if the last viral load within the Week 24 visit window was <50/c/mL, regardless of the ART regimen they were on at the time of viral load assessment (in other words switch from DTG plus 3TC fixed-dose combination [FDC] to another ART was not penalized) and as HIV-1 RNA >= 50 c/mL in all other cases (i.e. last viral load within Week 24 visit window >= 50 c/mL, on study but having missing viral load data at Week 24, discontinued early from study due to lost to follow-up (LFU), withdrew consent or any other reason). Confidence intervals (CI) were calculated based on the Exact Clopper-Pearson method. Percentage of participants with plasma HIV-1 RNA < 50 c/mL based on ITT-E missing = Failure analysis at Week 24 are presented.
Time Frame: At Week 24
Population: Intent-To-Treat Exposed (ITT-E) Population was used which comprised of all enrolled participants who received at least one dose of study treatment. ITT-E missing = Failure analysis is mentioned as 'Observed analysis' in the protocol.
Measure: Number (95% Confidence Interval); unit: Percentage of Participants
Arm/Group | DTG Plus 3TC
Number analyzed (Participants) | 131
Percentage of Participants | 78 [69.8 to 84.6]

2. Secondary Outcome: Percentage of Participants With Plasma HIV-1 RNA <50 c/mL Regardless of ART Regimen at Week 48 by ITT-E Missing = Failure Analysis
Description: Participants were classified as "HIV-1 RNA <50 c/mL" using an ITT-E Missing = Failure analysis. Participants were classified as 'HIV-1 RNA < 50 c/mL' if the last viral load within the Week 48 visit window was <50/c/mL, regardless of the ART regimen they were on at the time of viral load assessment (in other words switch from DTG plus 3TC FDC to another ART was not penalized) and as HIV-1 RNA >= 50 c/mL in all other cases (i.e. last viral load within Week 48 visit window >= 50 c/mL, on study but having missing viral load data at Week 48, discontinued early from study due to LFU, withdrew consent or any other reason). CI were calculated based on the Exact Clopper-Pearson method. Percentage of participants with plasma HIV-1 RNA < 50 c/mL based on ITT-E missing = Failure analysis at Week 48 are presented.
Time Frame: At Week 48
Population: Intent-to-Treat Exposed Population
Measure: Number (95% Confidence Interval); unit: Percentage of Participants
Arm/Group | DTG Plus 3TC
Number analyzed (Participants) | 131
Percentage of Participants | 82 [74.0 to 87.9]

3. Other Pre Specified Outcome: Percentage of Participants With HIV-1 RNA < 50 c/mL at Weeks 24 and 48 Among Participants With Available HIV-1 RNA Assessment Regardless of ART
Description: Participants with at least one viral load assessment within Week 24 and 48 visit window have been considered. Participants who discontinued from study prior to Week 24 and Week 48 or who were still on study at Week 24 and Week 48 but with missing viral load assessment have been excluded. Viral load assessments performed under DTG + 3TC FDC treatment or under any Modified ART treatment at Week 24 and Week 48 have been considered. Percentage of participants with HIV-1 RNA < 50 c/mL at Weeks 24 and 48 among participants with available HIV-1 RNA assessment regardless of ART have been presented.
Time Frame: At Week 24 and Week 48
Population: Intent-to-Treat Exposed Population. Only those participants with data available at the specified time points were analyzed (represented by n=X in the category titles).
Measure: Number; unit: Percentage of Participants
Arm/Group | DTG Plus 3TC
Number analyzed (Participants) | 111
Percentage of Participants
  Week 24, n=111 | 92
  Week 48, n=110: number analyzed (Participants) | 110
  Week 48, n=110 | 97

4. Secondary Outcome: Percentage of Participants With Plasma HIV-1 RNA <50 c/mL Using Food and Drug Administration (FDA) Snapshot Algorithm
Description: Percentage of participants with HIV-1 RNA<50 c/mL was obtained using FDA Snapshot algorithm. The Snapshot algorithm treated all participants without HIV-1 RNA data at the visit of interest (either due to missing plasma HIV-1 RNA assessment but on study, or due to permanent discontinuation of study treatment prior to visit window) as virologic non-success, as well as participants who switched from first line regimen of DTG + 3TC FDC for any reason prior to the visit of interest. Confidence intervals were calculated based on the Exact Clopper-Pearson method. Percentage of participants with plasma HIV-1 RNA <50 c/mL obtained using FDA Snapshot algorithm are presented.
Time Frame: At Week 24 and Week 48
Population: Intent-to-Treat Exposed Population
Measure: Number (95% Confidence Interval); unit: Percentage of Participants
Arm/Group | DTG Plus 3TC
Number analyzed (Participants) | 131
Percentage of Participants
  Week 24 | 74 [65.7 to 81.3]
  Week 48 | 76 [68.1 to 83.3]

5. Secondary Outcome: Time to Viral Suppression (HIV-1 RNA<50 c/mL) for Participants Who Had HIV-1 RNA >= 50 c/mL at Baseline
Description: Time of viral suppression for participants who had HIV-1 RNA >= 50 c/mL at Baseline is defined as the time to first viral load value < 50 c/mL, irrespective of the ART regimen a participant was on when that occurred. Non parametric Kaplan-Meier method was used. Participants who withdrew for any reason without being suppressed were censored at date of withdrawal. Participants who have not been withdrawn and have not had viral suppression at time of the analysis were censored at last viral load date. Median time (i.e. time when 50% of participants have reached HIV-1 RNA < 50 c/mL) along with 95% CI is presented.
Time Frame: Up to Week 48
Population: Intent-to-Treat Exposed Population. Only those participants with data available at the specified time points were analyzed.
Measure: Median (95% Confidence Interval); unit: Days
Arm/Group | DTG Plus 3TC
Number analyzed (Participants) | 126
Days | 35 [30 to 55]

6. Secondary Outcome: Number of Participants Who Changed First Line Regimen of DTG + 3TC FDC Due to Baseline Laboratory Results or HIV-1 Resistance Mutation Results
Description: Number of participants who switched from first line regimen of DTG + 3TC FDC due to abnormal Baseline laboratory values or Baseline HIV-1 resistance mutation results are presented.
Time Frame: Up to Week 48
Population: Intent-to-Treat Exposed Population
Measure: Count of Participants; unit: Participants
Arm/Group | DTG Plus 3TC
Number analyzed (Participants) | 131
Participants
  Switched due to abnormal Baseline laboratory results (HBV Infection) | 5
  Switched due to HIV-1 resistance mutation results | 1

7. Secondary Outcome: Number of Participants With Treatment-emergent Genotypic Resistance
Description: Blood samples were collected for genotypic resistance testing post-Baseline when Confirmed Virologic Failure criteria were met or in other occasion as needed (e.g. at time of study withdrawal when HIV-1 RNA >= 400 c/mL). New mutations were tabulated by drug class: integrase strand transfer inhibitor (INSTI), non-nucleoside reverse transcriptase inhibitor (NNRTI), nucleoside reverse transcriptase inhibitor (NRTI) and protease inhibitor (PI). Number of participants with treatment-emergent resistance associated mutations to any class (INSTI, NNRTI, NRTI, PI) from post-Baseline genotypic resistance data up to Week 48 have been presented.
Time Frame: Up to Week 48
Population: HIV-1 Viral Genotypic Population comprised of all participants in the ITT-E Population who had available post-Baseline HIV-1 genotypic resistance data either for DTG + 3TC FDC or any other ART. Only those participants with data available at the specified time points were analyzed.
Measure: Count of Participants; unit: Participants
Arm/Group | DTG Plus 3TC
Number analyzed (Participants) | 4
Participants
  NNRTI | 0
  INSTI | 0
  NRTI | 0
  PI | 0

8. Secondary Outcome: Number of Participants With Treatment-emergent Phenotypic Resistance
Description: Blood samples were collected for drug resistance testing post-Baseline when Confirmed Virologic Failure criteria were met or in other occasion as needed (e.g. at time of study withdrawal when HIV-1 RNA >= 400 c/mL). Assessment of antiviral activity of ART using phenotypic test results was interpreted through a proprietary algorithm (from Monogram Biosciences) and provides the overall susceptibility of the drug. Number of participants with phenotypic resistance to DTG and/or 3TC or any other ART (if treatment is modified) taken during the study in participants with post-Baseline phenotypic resistance data up to Week 48 have been presented.
Time Frame: Up to Week 48
Population: HIV-1 Viral Phenotypic Population comprised of all participants in the ITT-E Population who had available post-Baseline HIV-1 phenotypic resistance data either under treatment with DTG + 3TC FDC or any other ART. Only those participants with data available at the specified time points were analyzed.
Measure: Count of Participants; unit: Participants
Arm/Group | DTG Plus 3TC
Number analyzed (Participants) | 3
Participants | 0

9. Secondary Outcome: Number of Participants With Any Serious Adverse Events (SAEs) and Any Common (>=2%) Non-serious Adverse Events (Non-SAEs) Under Treatment With DTG + 3TC FDC
Description: An adverse event is any untoward medical occurrence in a clinical study participant, temporally associated with the use of a medicinal product, whether or not considered related to the medicinal product. An SAE is defined as any untoward medical occurrence that; results in death, is life-threatening, requires hospitalization or prolongation of existing hospitalization, results in disability/incapacity, is a congenital anomaly/birth defect, other situations as judged by physician. Number of participants with any SAE and common (>=2%) non-SAEs are presented.
Time Frame: Up to Week 48
Population: Safety Population comprised of all enrolled participants who received at least one dose of study treatment.
Measure: Count of Participants; unit: Participants
Arm/Group | DTG Plus 3TC
Number analyzed (Participants) | 131
Participants
  Any non-SAE | 85
  Any SAE | 2

10. Secondary Outcome: Number of Participants With Maximum Post-Baseline Emergent Hematology Toxicities Under Treatment With DTG + 3TC FDC
Description: Blood samples were collected up to Week 48 visit for the analysis of hematology parameters-platelet count, neutrophils, hemoglobin and leukocytes Any abnormality was graded according to Division of Acquired Immunodeficiency Syndrome (DAIDS) toxicity scales from Grade 1 to 4 (1=Mild, 2=Moderate, 3=Severe, 4=Potentially life threatening). Higher grade indicates more severity. Only those participants with maximum post-Baseline emergent hematology toxicities in any of the hematology parameters have been presented.
Time Frame: Up to Week 48
Population: Safety Population
Measure: Count of Participants; unit: Participants
Arm/Group | DTG Plus 3TC
Number analyzed (Participants) | 131
Participants
  Hemoglobin, Grade 1 | 5
  Hemoglobin, Grade 2 | 1
  Hemoglobin, Grade 3 | 0
  Hemoglobin, Grade 4 | 0
  Leukocytes, Grade 1 | 5
  Leukocytes, Grade 2 | 2
  Leukocytes, Grade 3 | 1
  Leukocytes, Grade 4 | 0
  Neutrophils, Grade 1 | 4
  Neutrophils, Grade 2 | 4
  Neutrophils, Grade 3 | 2
  Neutrophils, Grade 4 | 1
  Platelets, Grade 1 | 1
  Platelets, Grade 2 | 1
  Platelets, Grade 3 | 0
  Platelets, Grade 4 | 0

11. Secondary Outcome: Number of Participants With Maximum Post-Baseline Emergent Chemistry Toxicities Under Treatment With DTG + 3TC FDC
Description: Blood samples were collected up to Week 48 for the analysis of clinical chemistry parameters: alanine aminotransferase (ALT), albumin, aspartate aminotransferase (AST), Alkaline Phosphatase (ALP), bilirubin, carbon dioxide (CO2), creatinine kinase (CK), creatinine, glomerular filtration rate (GFR) from creatinine adjusted for body surface area (BSA), glucose, hypercalcemia, hyperkalemia, hypernatremia, hypocalcemia, hypokalemia, hyponatremia and phosphate. Any abnormality was graded according to DAIDS toxicity scales from Grade 1 to 4 (1=Mild, 2=Moderate, 3=Severe, 4=Potentially life threatening). Higher grade indicates more severity. Only those participants with maximum post-Baseline emergent chemistry toxicities in any of the chemistry parameters have been presented.
Time Frame: Up to Week 48
Population: Safety Population
Measure: Count of Participants; unit: Participants
Arm/Group | DTG Plus 3TC
Number analyzed (Participants) | 131
Participants
  ALT, Grade 1 | 7
  ALT, Grade 2 | 2
  ALT, Grade 3 | 0
  ALT, Grade 4 | 1
  Albumin, Grade 1 | 0
  Albumin, Grade 2 | 1
  Albumin, Grade 3 | 0
  Albumin, Grade 4 | 0
  AST, Grade 1 | 6
  AST, Grade 2 | 1
  AST, Grade 3 | 1
  AST, Grade 4 | 1
  Bilirubin, Grade 1 | 5
  Bilirubin, Grade 2 | 0
  Bilirubin, Grade 3 | 1
  Bilirubin, Grade 4 | 0
  CO2, Grade 1 | 20
  CO2, Grade 2 | 0
  CO2, Grade 3 | 0
  CO2, Grade 4 | 0
  CK, Grade 1 | 0
  CK, Grade 2 | 1
  CK, Grade 3 | 0
  CK, Grade 4 | 0
  Creatinine, Grade 1 | 9
  Creatinine, Grade 2 | 1
  Creatinine, Grade 3 | 2
  Creatinine, Grade 4 | 0
  GFR from creatinine adjusted for BSA,Grade 1 | 0
  GFR from creatinine adjusted for BSA,Grade 2 | 38
  GFR from creatinine adjusted for BSA,Grade 3 | 8
  GFR from creatinine adjusted for BSA,Grade 4 | 1
  Glucose, Grade 1 | 27
  Glucose, Grade 2 | 14
  Glucose, Grade 3 | 2
  Glucose, Grade 4 | 0
  Hypercalcaemia, Grade 1 | 5
  Hypercalcaemia, Grade 2 | 0
  Hypercalcaemia, Grade 3 | 0
  Hypercalcaemia, Grade 4 | 0
  Hyperkalemia, Grade 1 | 0
  Hyperkalemia, Grade 2 | 1
  Hyperkalemia, Grade 3 | 0
  Hyperkalemia, Grade 4 | 0
  Hypernatremia, Grade 1 | 2
  Hypernatremia, Grade 2 | 0
  Hypernatremia, Grade 3 | 0
  Hypernatremia, Grade 4 | 0
  Hypokalemia, Grade 1 | 1
  Hypokalemia, Grade 2 | 0
  Hypokalemia, Grade 3 | 0
  Hypokalemia, Grade 4 | 0
  Hyponatremia, Grade 1 | 9
  Hyponatremia, Grade 2 | 0
  Hyponatremia, Grade 3 | 0
  Hyponatremia, Grade 4 | 0
  Phosphate, Grade 1 | 8
  Phosphate, Grade 2 | 0
  Phosphate, Grade 3 | 0
  Phosphate, Grade 4 | 0
  Hypocalcaemia, Grade 1 | 5
  Hypocalcaemia, Grade 2 | 1
  Hypocalcaemia, Grade 3 | 0
  Hypocalcaemia, Grade 4 | 0
  ALP, Grade 1 | 1
  ALP, Grade 2 | 0
  ALP, Grade 3 | 0
  ALP, Grade 4 | 0

12. Secondary Outcome: Number of Participants Who Discontinued the Study Treatment (DTG+3TC FDC) Due to AEs
Description: An adverse event is any untoward medical occurrence in a clinical study participant, temporally associated with the use of a medicinal product, whether or not considered related to the medicinal product. Number of participants who discontinued the study treatment (DTG plus 3TC) due to AEs are presented.
Time Frame: Up to Week 48
Population: Safety Population
Measure: Count of Participants; unit: Participants
Arm/Group | DTG Plus 3TC
Number analyzed (Participants) | 131
Participants | 1

13. Secondary Outcome: Number of Participants Who Discontinued the Study Treatment (DTG+3TC FDC) Due to Drug-related AEs
Description: An adverse event is any untoward medical occurrence in a clinical study participant, temporally associated with the use of a medicinal product, whether or not considered related to the medicinal product. Number of participants who discontinued the study treatment (DTG+3TC FDC) due to drug-related AEs are presented.
Time Frame: Up to Week 48
Population: Safety Population
Measure: Count of Participants; unit: Participants
Arm/Group | DTG Plus 3TC
Number analyzed (Participants) | 131
Participants | 1

14. Secondary Outcome: Change From Baseline in Cluster of Differentiation (CD4+) Cell Counts for Participants Under Treatment With DTG + 3TC FDC
Description: CD4+ cells are type of white blood cells that fight infection and as HIV infection progresses, the number of these cells decline. Blood samples were collected at specified time points to assess CD4+. It was evaluated by flow cytometry. Baseline value is defined as the latest pre-dose assessment (Day 1). Change from Baseline was defined as post-dose visit value minus Baseline value.
Time Frame: Baseline (Day 1) and Week 24 and Week 48
Population: as for outcome 3
Measure: Mean (Standard Deviation); unit: Cells per cubic millimeter
Arm/Group | DTG Plus 3TC
Number analyzed (Participants) | 106
Cells per cubic millimeter
  Week 24, n=106 | 185.9 (163.70)
  Week 48, n=103: number analyzed (Participants) | 103
  Week 48, n=103 | 273.4 (223.93)

15. Secondary Outcome: Change From Baseline in CD4+/CD8+ Cell Count Ratio for Participants Under Treatment With DTG + 3TC FDC
Description: Blood samples were collected at specified time points to assess CD4+/CD8+ cell count ratio. It was assessed by flow cyclometry to evaluate the immunologic activity of DTG plus 3TC. Baseline value is defined as the latest pre-dose assessment (Day 1). Change from Baseline was defined as post-dose visit value minus Baseline value.
Time Frame: Baseline (Day 1) and Week 24 and Week 48
Population: as for outcome 3
Measure: Mean (Standard Deviation); unit: Ratio
Arm/Group | DTG Plus 3TC
Number analyzed (Participants) | 106
Ratio
  Week 24, n= 106 | 0.30 (0.238)
  Week 48, n=102: number analyzed (Participants) | 102
  Week 48, n=102 | 0.39 (0.260)

16. Secondary Outcome: Number of Participants With HIV-1 Disease Progression to Stage 3 HIV-associated Conditions, Acquired Immunodeficiency Syndrome (AIDS) or Death (for Participants Under Treatment With DTG + 3TC FDC)
Description: HIV-associated conditions were recorded during the study and was assessed according to the 2014 Centers for Disease Control and Prevention (CDC) Classification System for HIV Infection in Adults. CDC classification for HIV were stage 1, 2 and 3. Higher stage indicates more severity. Disease progression summarize participants who had HIV infection stage 3 associated conditions, AIDS and/or death. Number of participants with HIV-1 disease progression to stage 3 HIV-associated conditions, AIDS or death are presented.
Time Frame: Up to Week 48
Population: Intent-to-Treat Exposed Population
Measure: Count of Participants; unit: Participants
Arm/Group | DTG Plus 3TC
Number analyzed (Participants) | 131
Participants | 1

17. Secondary Outcome: Number of Participants Who Completed 24 and 48 Weeks on Study
Description: Number of participants who completed 24 and 48 weeks on study are presented.
Time Frame: Week 24 and Week 48
Population: Intent-to-Treat Exposed Population
Measure: Count of Participants; unit: Participants
Arm/Group | DTG Plus 3TC
Number analyzed (Participants) | 131
Participants
  Week 24 | 115
  Week 48 | 112

18. Secondary Outcome: Number of Participants Retained in Care for 24 and 48 Weeks on Study and Have HIV-1 RNA <200 c/mL
Description: Number of participants retained in care for 24 and 48 weeks on study and have HIV-1 RNA <200 c/mL have been presented.
Time Frame: Week 24 and Week 48
Population: Intent-to-Treat Exposed Population
Measure: Count of Participants; unit: Participants
Arm/Group | DTG Plus 3TC
Number analyzed (Participants) | 131
Participants
  Week 24 | 110
  Week 48 | 109

ADVERSE EVENTS:
Time Frame: Serious adverse events (SAEs) and non-serious adverse events were collected from start of study treatment (Week 1) up to end of the study (Week 48).
Description: SAEs and non-serious adverse events were reported for the Safety Population which comprised of all enrolled participants who received at least one dose of study treatment.
Arm/Group | DTG Plus 3TC
All-Cause Mortality (participants affected / at risk) | 0/131
Serious Adverse Events (participants affected / at risk) | 2/131
Other Adverse Events (participants affected / at risk) | 85/131
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | DTG Plus 3TC (N=131)
Cellulitis (Infections and infestations) | 1
Streptococcal bacteraemia (Infections and infestations) | 1
OTHER ADVERSE EVENTS (reported when occurring in more than 2% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | DTG Plus 3TC (N=131)
Diarrhoea (Gastrointestinal disorders) | 11
Nausea (Gastrointestinal disorders) | 9
Abdominal discomfort (Gastrointestinal disorders) | 3
Constipation (Gastrointestinal disorders) | 5
Headache (Nervous system disorders) | 12
Dizziness (Nervous system disorders) | 5
Paraesthesia (Nervous system disorders) | 3
Nasopharyngitis (Infections and infestations) | 8
Chlamydial infection (Infections and infestations) | 4
Gonorrhoea (Infections and infestations) | 5
Upper respiratory tract infection (Infections and infestations) | 3
Pruritus (Skin and subcutaneous tissue disorders) | 7
Rash (Skin and subcutaneous tissue disorders) | 8
Acne (Skin and subcutaneous tissue disorders) | 3
Insomnia (Psychiatric disorders) | 8
Depression (Psychiatric disorders) | 9
Fatigue (General disorders) | 8
Pyrexia (General disorders) | 4
Weight increased (Investigations) | 8
Exposure to communicable disease (Injury, poisoning and procedural complications) | 6
Neck pain (Musculoskeletal and connective tissue disorders) | 3
Cough (Respiratory, thoracic and mediastinal disorders) | 4
Hypertension (Vascular disorders) | 5
Anogenital dysplasia (Gastrointestinal disorders) | 4
Anxiety (Psychiatric disorders) | 7
COVID-19 (Infections and infestations) | 5
Proctitis gonococcal (Infections and infestations) | 4
Anal chlamydia infection (Infections and infestations) | 3
Herpes simplex (Infections and infestations) | 3
Herpes zoster (Infections and infestations) | 3
Oropharyngeal gonococcal infection (Infections and infestations) | 3
Pharyngitis (Infections and infestations) | 3
Tonsillitis (Infections and infestations) | 3
Arthralgia (Musculoskeletal and connective tissue disorders) | 6
Pain in extremity (Musculoskeletal and connective tissue disorders) | 3
Anogenital warts (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 4
Vitamin D deficiency (Metabolism and nutrition disorders) | 3
Haemorrhoids (Gastrointestinal disorders) | 4

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
GSK agreements may vary with individual investigators, but will not prohibit any investigator from publishing. GSK supports the publication of results from all centers of a multi-center trial but requests that reports based on single-site data not precede the primary publication of the entire clinical trial.

DOCUMENTS (2):
  • Study Protocol (2019-06-06): https://cdn.clinicaltrials.gov/large-docs/81/NCT03945981/Prot_000.pdf
  • Statistical Analysis Plan (2019-06-20): https://cdn.clinicaltrials.gov/large-docs/81/NCT03945981/SAP_001.pdf